CLINICAL TRIAL: NCT01556321
Title: Long-term Effects of Green Tea on Gut Flora, Fat Absorption, Body Composition and Resting Energy Expenditure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NL38773
Record Dates: First submitted 2012-03-07; First posted 2012-03-16 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2013-05

CONDITIONS: Obesity
Keywords: Obesity; Body weight; Gut flora; Fat absorption
MeSH Terms: conditions — Obesity; Body Weight | interventions — Tea; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Green tea, normal weight (Experimental): Subjects with a BMI 18.5-25 kg/m2 will receive green tea capsules, which they have to consume daily for a period of twelve weeks
  Interventions: Dietary Supplement: green tea (757 mg/capsule [84.5 mg EGCG + 2.1 mg caffeine ]
- Placebo, normal weight (Placebo Comparator): Subjects with a BMI 18.5-25 kg/m2 will receive placebo capsules, which they have to consume daily for a period of twelve weeks
  Interventions: Dietary Supplement: placebo
- Green tea, overweight (Experimental): Subjects with a BMI >30 kg/m2 will receive green tea capsules, which they have to consume daily for a period of twelve weeks
  Interventions: Dietary Supplement: green tea (757 mg/capsule [84.5 mg EGCG + 2.1 mg caffeine ]
- Placebo capsules, obese (Placebo Comparator): Subjects with a BMI >30 kg/m2 will receive placebo capsules, which they have to consume daily for a period of twelve weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: placebo — Subjects will receive placebo (soy oil; 757 mg/capsule, 3 capsules with each breakfast, lunch and dinner) in capsule form after their baseline measurement, which they have to consume daily for a period of twelve weeks.
  Arms: Placebo capsules, obese; Placebo, normal weight
Dietary Supplement: green tea (757 mg/capsule [84.5 mg EGCG + 2.1 mg caffeine ] — Subjects will receive green tea (757 mg/capsule [84.5 mg EGCG + 2.1 mg caffeine ], 3 capsules with each breakfast, lunch and dinner)in capsule form after their baseline measurement, which they have to consume daily for a period of twelve weeks.
  Arms: Green tea, normal weight; Green tea, overweight

SUMMARY:
Green tea may have positive effects for weight control and on body composition via several approaches such as a positive effect on the gut flora, a decrease in fat absorption from the intestines and an increase in resting energy expenditure.

DETAILED DESCRIPTION:
Green tea may have positive effects for weight control and on body composition via several approaches such as a positive effect on the gut flora, a decrease in fat absorption from the intestines and an increase in resting energy expenditure. We would like to investigate the long-term effects of green tea on gut flora, fat absorption, resting energy expenditure and body composition.

The study will be conducted in a randomized, placebo-controlled, double-blind parallel design with four groups consisting of control groups and green tea groups with normal weight subjects and obese subjects. At three time points (baseline, 6 weeks and 12 weeks) faeces are collected for analyzing the gut flora composition and fat content. Furthermore, measurements of resting energy expenditure and body composition will be conducted. Activity will be measured during three weeks (baseline, week 6 and week 12).

a hundred healthy subjects (50 males and 50 females) with a BMI between 18.5-25 kg/m2 and ≥30 kg/m2 and aged between 18-50 years will be included in the study. All subjects will be non-smoking, non tea-drinkers, weight stable, dietary unrestraint, and at most moderate alcohol and caffeine consumers. Subjects will be free of medication except for oral contraceptives use in women.

Intervention (if applicable):

Subjects will receive either green tea or placebo in capsule form after their baseline measurement, which they have to consume three times daily for a period of twelve weeks.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.5-25 kg/m2 and ≥30 kg/m2
* Age between 18-50 years
* Healthy
* Weight stable
* Dietary unrestraint
* Not using a more than moderate amount of alcohol (>10 consumptions/wk)
* Not using more than 100 mg caffeine per day
* Not drinking tea
* Not using probiotics
* Being weight stable (weight change < 3kg during the last 6 months)
* Dietary unrestraint
* Not using antibiotics during the last 6 months.
* Free of medication except for oral contraceptives use in women.

Exclusion Criteria:

* Not healthy
* Smoking
* Using a more than moderate amount of alcohol
* Using more than 100 mg caffeine per day
* Drinking tea
* Using probiotics
* Not being weight stable
* Dietary restraint
* Using medication or supplements except for oral contraceptives in women
* Using antibiotics
* Not meeting the criteria for BMI and age.
* Pregnant or lactating women
* Having allergies for the used food items will also be excluded from participation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2012-06; Primary Completion 2014-12 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Faeces are collected for analyzing the gut flora and fat absorption | At three time points (baseline, 6 weeks and 12 weeks)
  The primary endpoint of this study is the change in gut flora; ratio firmicutes/bacteroidetes, changes in total faecal fat and change in body weight.

SECONDARY OUTCOMES:
Resting energy expenditure (REE) | At three time points (baseline, 6 weeks and 12 weeks)
Respiratory quotient (RQ) | At three time points (baseline, 6 weeks and 12 weeks)
Three frequency eating questionnaire (TFEQ) | At three time points (baseline, 6 weeks and 12 weeks)
Body composition: BMI, body fat percentage, fat mass index (FMI) | At three time points (baseline, 6 weeks and 12 weeks)
Body fat distribution: waist circumference, waist-to-hip ratio (WHR | At three time points (baseline, 6 weeks and 12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Margriet Westerterp-Plantenga, Prof. Dr., Principal Investigator — Maastricht University, department of human biology
Locations (1):
- Maastricht University, Human Biology, Maastricht, Netherlands

REFERENCES:
- [Background] Hursel R, Viechtbauer W, Dulloo AG, Tremblay A, Tappy L, Rumpler W, Westerterp-Plantenga MS. The effects of catechin rich teas and caffeine on energy expenditure and fat oxidation: a meta-analysis. Obes Rev. 2011 Jul;12(7):e573-81. doi: 10.1111/j.1467-789X.2011.00862.x. Epub 2011 Mar 2. PMID 21366839
- [Background] Hursel R, Viechtbauer W, Westerterp-Plantenga MS. The effects of green tea on weight loss and weight maintenance: a meta-analysis. Int J Obes (Lond). 2009 Sep;33(9):956-61. doi: 10.1038/ijo.2009.135. Epub 2009 Jul 14. PMID 19597519
- [Derived] Janssens PL, Penders J, Hursel R, Budding AE, Savelkoul PH, Westerterp-Plantenga MS. Long-Term Green Tea Supplementation Does Not Change the Human Gut Microbiota. PLoS One. 2016 Apr 7;11(4):e0153134. doi: 10.1371/journal.pone.0153134. eCollection 2016. PMID 27054321
- [Derived] Janssens PL, Hursel R, Westerterp-Plantenga MS. Long-term green tea extract supplementation does not affect fat absorption, resting energy expenditure, and body composition in adults. J Nutr. 2015 May;145(5):864-70. doi: 10.3945/jn.114.207829. Epub 2015 Mar 4. PMID 25740906